CLINICAL TRIAL: NCT02532647
Title: A Study Evaluating the Safety and Efficacy of Remimazolam (CNS 7056) Compared to Placebo and Midazolam in ASA III and IV Patients Undergoing Colonoscopy
Brief Title: Safety and Efficacy of Remimazolam in ASA III and IV Patients Undergoing Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CNS7056-015
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Experimental): Remimazolam 2.5 - 5.0 mg initially, followed by 1.25 - 2.5 mg top-up doses as required to maintain sedation.
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Remimazolam
- Midazolam (Active Comparator): Midazolam 1.0 mg initially, followed by 0.5 mg top-up doses as required to maintain sedation.
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Midazolam
- Placebo (Placebo Comparator): Placebo administered in double-blind manner.
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remimazolam
  Other Names: CNS7056
  Arms: Remimazolam
Drug: Midazolam
  Other Names: Versed
  Arms: Midazolam
Drug: Placebo
  Arms: Placebo

SUMMARY:
A prospective, double-blind, randomized, placebo and active controlled, multi-center, parallel group study comparing remimazolam to placebo, with an additional open-label arm for midazolam, in American Society of Anesthesiologists (ASA) Grade III and IV patients (ASA status evaluated by an anesthesiologist not otherwise involved in the study) undergoing a colonoscopy for diagnostic or therapeutic reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged ≥18, scheduled to undergo a diagnostic or therapeutic colonoscopy (therapeutic procedures may include hemostasis, resection, ablation decompression, and foreign body extraction, for example).
2. ASA grade III/IV

   1. ASA III patients are patients with severe systemic disease eg patients who, in the judgment of the Principal Investigator (PI), have significant enough systemic disease to warrant performing the colonoscopy procedure only in a facility which has post-procedure inpatient capability. ASA III physical status classification encompasses a wide range of potential patient co-morbidities some of which may make the selection of a facility with post-procedure inpatient capability preferable. By definition, ASA III patients have one or more moderate to severe systemic diseases which potentially cause substantial functional limitation. Examples may include poorly controlled diabetes or hypertension, moderate to severe chronic obstructive pulmonary disease, active hepatitis, heart failure or coronary artery disease (including implanted pacemaker and/or stent, recent myocardial infarction) cerebrovascular accident, or end stage renal disease requiring dialysis.
   2. ASA IV patients are patients with severe systemic disease that is a constant threat to life eg at least one severe disease that is poorly controlled or at end stage; possible risk of death; unstable angina; symptomatic chronic obstructive pulmonary disease; symptomatic chronic heart failure; hepatorenal failure.
3. For all female patients, negative result of urine or serum pregnancy test. Additionally, for women with child-bearing potential only, use of birth control during the study period (from the time of consent until all specified observations are completed).
4. Patient voluntarily signs and dates an informed consent form (ICF) that is approved by an investigational review board (IRB) prior to the conduct of any study procedure.
5. Patient is willing and able to comply with study requirements and will be available for a Follow-up Visit on Day 1 (+ 1 day) and Follow-up Phone call (Day 4 +/- 3 days) after the colonoscopy.

Exclusion Criteria:

1. Patients with a known sensitivity to benzodiazepines, flumazenil, opioids, naloxone, or a medical condition such that these agents are contraindicated.
2. Female patients with a positive pregnancy test at screening or baseline and lactating female patients.
3. Patients clearly acutely intoxicated with alcohol or drugs of abuse at baseline.
4. Patients in receipt of any investigational drug within 30 days or less than 7 half-lives (whichever is longer) before Screening, or scheduled to receive one during the study period.
5. Participation in any previous clinical trial with remimazolam.
6. Patients with an inability to communicate well with the Investigator, or deemed unsuitable according to the Investigator (in each case providing a reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, MD, Principal Investigator — IU Health University Hospital
Locations (3):
- United States (3):
  - Jupiter Medical Center, Jupiter, Florida
  - Indiana University Division of Gastroenterology/Hepatology, Indianapolis, Indiana
  - Delta Research Partners Inc, Monroe, Louisiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Remimazolam: Remimazolam 2.5 - 5.0 mg initially, followed by 1.25 - 2.5 mg top-up doses as required to maintain sedation.
- Placebo: Placebo administered in double-blind manner.
- Midazolam: Midazolam 1.0 mg initially, followed by 0.5 mg top-up doses as required to maintain sedation.
Period: Overall Study
Arm/Group | Remimazolam | Placebo | Midazolam
Started | 32 | 16 | 31
Safety Population (Safety Population: all randomised patients who received any amount of trial drug) | 31 | 16 | 30
Completed | 31 | 16 | 30
Not Completed | 1 | 0 | 1
Not completed — Did not receive trial medication | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Remimazolam | Placebo | Midazolam | Total
Number analyzed (Participants) | 31 | 16 | 30 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.65) | 63.0 (8.37) | 61.5 (10.60) | 62.5 (9.32)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 18 | 9 | 19 | 46
  ≥65 years | 13 | 7 | 11 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 16 | 34
  Male | 17 | 12 | 14 | 43
Region of Enrollment [Number; unit: participants]
  United States | 31 | 16 | 30 | 77
Height [Mean (Standard Deviation); unit: cm] | 171.1 (10.07) | 171.8 (7.72) | 168.4 (10.32) | 170.2 (9.72)
Weight [Mean (Standard Deviation); unit: kg] | 91.0 (28.14) | 94.0 (26.11) | 87.9 (23.91) | 90.4 (25.90)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 30.9 (8.28) | 30.8 (5.53) | 30.8 (6.75) | 30.8 (7.11)
American Society of Anesthesiologists (ASA) Classification [Count of Participants; unit: Participants] — ASA Class III: Severe systemic disease. ASA Class IV: Severe systemic disease that is constant threat to life
  Participants
    ASA Class III | 16 | 9 | 15 | 40
    ASA Class IV | 15 | 7 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Success Rates of the Procedure
Description: The success of the procedure, as measured by completion of the colonoscopy procedure, AND no requirement for a rescue sedative medication, AND no requirement of more than 5 doses of study medication within any 15 minute window. (For midazolam: 3 doses within any 12 minute window)
Time Frame: From first dose of study drug until the end of colonoscopy
Population: All patients who were randomised, and analysed as randomised.
Measure: Count of Participants; unit: Participants
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 32 | 16 | 31
Participants | 27 | 0 | 4

2. Secondary Outcome: Time to Start of Procedure
Description: The time from the first administration of the study drug to the beginning of the colonoscopy
Time Frame: From the first administration of the study drug to the beginning of the colonoscopy
Population: Patients who did not reach the endpoint are excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 31 | 16 | 30
minutes | 5.0 [4.0 to 8.0] | 18.3 [17.5 to 21.0] | 19.0 [19.0 to 19.0]

3. Secondary Outcome: Time to Fully Alert
Description: Time to first of 3 Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores of 5 after the end of colonoscopy procedure (colonoscope out) and after the last injection of study drug
Time Frame: From the last injection of the study drug AND from end of colonoscopy until the patient has recovered to fully alert
Population: Patients who did not reach the endpoint are censored at last observation.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 31 | 16 | 30
minutes
  After last dose of trial or rescue sedative | 11.0 [8.8 to 12.0] | 18.0 [14.0 to 25.0] | 18.8 [15.0 to 26.0]
  After the end of colonoscopy | 3.0 [2.0 to 4.0] | 5.3 [4.0 to 12.0] | 7.0 [4.0 to 12.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected from first dose of study drug medication until Day 4 (+ 3 days), and were followed until events resolved, became stable, or could be explained by another known cause(s)
Description: Total number of participants affected with Other (Not Including Serious) Adverse Events represents any participant in the trial with a TEAE. The number of participants with Preferred Term (PT)TEAEs represents participants with TEAEs reported with a threshold of 5% in any of the arms
Arm/Group | Remimazolam | Placebo | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/16 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/16 | 1/30
Other Adverse Events (participants affected / at risk) | 28/31 | 13/16 | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam (N=31) | Placebo (N=16) | Midazolam (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam (N=31) | Placebo (N=16) | Midazolam (N=30)
Hypotension (Vascular disorders) | 18 | 11 | 17
Hypertension (Vascular disorders) | 13 | 6 | 13
Diastolic hypertension (Vascular disorders) | 3 | 0 | 0
Diastolic hypotension (Vascular disorders) | 1 | 1 | 0
Systolic hypertension (Vascular disorders) | 2 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 8
Bradycardia (Cardiac disorders) | 1 | 1 | 4
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Respiratory rate decreased (Investigations) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 45 days prior to submission of communications, sponsor shall review and comment on the communications. Sponsor shall have the right to require institution and investigator to remove specifically identified confidential information and to delay the proposed publication an additional 45 days to enable sponsor to seek patent protection